CLINICAL TRIAL: NCT04877327
Title: X-TRA CLINICAL TRIAL (X-therapy for Redo AF Ablation). Strategy of Crossing Two Ablation Techniques (Cryoballoon and Radiofrequency) After the Recurrence of Paroxysmal AF and the Need for a New Procedure
Brief Title: Strategy of Crossing Two Ablation Techniques (Cryoballoon and Radiofrequency) After the Recurrence of Paroxysmal AF and the Need for a New Procedure
Acronym: X-TRA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low recruitment
Sponsor: Galaxia Empírica (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: X-TRA
Record Dates: First submitted 2021-04-28; First posted 2021-05-07 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cross-over of ablation technique (Experimental): Cross-over of cardiac ablation procedures (cryotherapy and radiofrequency; radiofrequency and cryotherapy)
  Interventions: Procedure: Ablation
- Repetition of the same technique (No Intervention): Repeat the same procedure (cryotherapy and cryotherapy; radiofrequency and radiofrequency)

INTERVENTIONS:
Procedure: Ablation — Cryotherapy and radiofrequency
  Arms: Cross-over of ablation technique

SUMMARY:
Randomized phase III clinical trial to compare the efficacy of the two most widely used ablation techniques (cryotherapy and radiofrequency) after recurrence of atrial fibrillation (AF) in patients requiring a new ablation procedure.

ELIGIBILITY:
Inclusion Criteria:

* Paroxysmal FA (one that ends, spontaneously or not, within 7 days of its onset. GUIDELINES ESC FA 2020)
* Have undergone an initial AF ablation procedure using Cryoballoon or point-to-point focal RF within the three years prior to the initial visit.
* During the initial AF ablation procedure ONLY pulmonary vein isolation / ablation will have been performed
* Documented recurrence of AF lasting more than 30 seconds after the first ablation procedure.
* With the ability and willingness to sign the informed consent of the patient.
* With a minimum follow-up capacity of 12 months.

Exclusion Criteria:

* Patients aged <18 years.
* Previous heart surgery.
* Moderate or severe mitral valve disease.
* Severe dilation of the left atrium, defined as a volume greater than 48 ml / m2 or a left atrial diameter greater than 50 mm in the parasternal long axis.
* Contraindication for anticoagulation.
* Pregnancy or pregnancy intention during the 12-month follow-up.
* Life expectancy less than 12 months.
* Unavailability for follow-up for 12 months.
* Simultaneous participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Compare the effectiveness of the technique crossover strategy versus the repetition of the same technique for the isolation of the pulmonary veins during a second ablation procedure indicated by recurrence of AF | 42 months
  The rate of recurrent AF will be documented to check whether it is better to cross ablation techniques or not.
  This efficacy is defined as the absence of documented AF recurrence lasting more than 30 seconds, during a 12-month follow-up after the second ablation procedure.

SECONDARY OUTCOMES:
To compare the efficacy of the AF re-ablation procedure based on the initial technique and the technique of the second procedure, during a 12-month follow-up after the second ablation procedure. | 42 months
  The patient's events during follow-up will be evaluated through follow-up visits and verification of his medical history and the rate of recurrent AF will be documented.
Analyze potential predictors of efficacy of each of the techniques based on the anatomy of the left atrium and pulmonary veins. Evaluate the number of reconnected pulmonary veins through cardiac imaging procedures | 42 months
  Evaluate the anatomical location of reconnection in each patient referred for re-ablation, depending on the technique used in the first procedure.

CONTACTS AND LOCATIONS:
Locations (9):
- Spain (9):
  - Hospital Universitario Virgen de las Nieves Granada, Granada, Andalusia
  - Hospital Virgen de la Victoria, Málaga, Andalusia
  - Complejo hospitalario universitario de Albacete, Albacete, Castille-La Mancha
  - Hospital Virgen de la Salud, Toledo, Castille-La Mancha
  - Complejo Hospitalario Universitario de Santiago de Compostela, Santiago de Compostela, Galicia
  - Hospital General Universitario de Alicante, Alicante, Valencia
  - Hospital Clínico Valencia, Valencia, Valencia
  - Hospital 12 de Octubre, Madrid
  - Hospital Puerta de Hierro, Madrid

IPD SHARING:
Plan to Share IPD: No